CLINICAL TRIAL: NCT04425655
Title: A Phase II Trial of Fludarabine in Combination With Daunorubicin and Cytarabine Liposome for Adults With Newly-diagnosed Acute Myeloid Leukemia: University of California Hematologic Malignancies Consortium Protocol 1914
Brief Title: Fludarabine in Combination With Daunorubicin and Cytarabine Liposome in Newly-diagnosed Acute Myeloid Leukemia.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Original investigator for the trial has left
Sponsor: University of California, San Diego (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, James Mangan, Associate Clinical Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCHMC1914
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Acute Myeloid Leukemia, Adult; AML; AML, Adult
Keywords: Vyxeos; CPX-351; Fludarabine; Untreated AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; fludarabine phosphate; CPX-351

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fludarabine and CPX351 (Experimental): Induction 1:
  Fludarabine 30 mg/m2/day IV on days 1-5 for 5 doses Daunorubicin and cytarabine liposome (CPX-351) daunorubicin 44 mg/m2/day and cytarabine 100 mg/m2/day IV on days 1, 3, 5 (given 4 hours after fludarabine infusion) for 3 doses
  Induction 2 (residual leukemia after Induction 1):
  Fludarabine 30 mg/m2/day IV on days 1-3 for 3 doses
  Daunorubicin and cytarabine liposome (CPX-351) daunorubicin 44 mg/m2/day and cytarabine 100 mg/m2/day IV on days 1, 3 (given 4 hours after fludarabine infusion) for 2 doses
  Optional consolidation, up to 2 cycles:
  Daunorubicin and cytarabine liposome (CPX-351) daunorubicin 29 mg/m2/day and cytarabine 65 mg/m2/day IV on days 1, 3 for 2 doses
  Interventions: Drug: Fludarabine; Drug: Vyxeos

INTERVENTIONS:
Drug: Fludarabine — 30mg/m2 days 1 through 5
  Other Names: Oforta, Fludara
Drug: Vyxeos — 100U/m2 days 1, 3 5 in induction, 65U/m2 days 1 and 3 for consolidation
  Other Names: CPX-351

SUMMARY:
This phase 2 clinical trial will evaluate the effectiveness and safety of fludarabine in combination with CPX-351 in patients with untreated AML. Patients will receive fludarabine and CPX-351 during Induction 1 and 2 as well as 2 cycles of consolidation therapy.

DETAILED DESCRIPTION:
This is a phase 2, open label single arm study to look at the effectives and safety of fludarabine in combination with CPX-351 in patients with untreated AML. The rationale for this combination stems from data which indicated that pre-treatment of the THP-1 cell line with fludarabine for 4 hours prior to CPX-351 administration (Flu-CPX) significantly potentiated intracellular ara-CTP accumulation compared to CPX-351 alone. This suggests that fludarabine combined with CPX-351 may have efficacy against leukemic clones that would be resistant to CPX-351 or standard chemotherapy in first induction. It has been demonstrated that treatment with CPX-351 produces superior clinical outcomes in secondary AML likely due to its novel formulation, which results in sustained exposure of the cytotoxic agents cytarabine and daunorubicin in a synergistic 5:1 ratio within the plasma and bone marrow. Fludarabine can potentially improve upon the outcomes observed with CPX-351 monotherapy and 7+3 by enhancing intracellular ara-CTP accumulation from CPX-351. Patients will received fludarabine and CPX-351 for up to 2 cycles of induction and 2 cycles of consolidation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed de novo or secondary AML as defined by WHO criteria
2. Intermediate- or poor-risk disease by ELN 2017 criteria
3. Adults 18 years of age or older
4. ECOG performance status of 0, 1, or 2
5. Able to give informed consent and follow study guidelines
6. Organ function requirements:

   1. Adequate renal function defined as creatinine clearance greater than 60 ml/min
   2. Adequate hepatic function defined by serum bilirubin less than or equal 2 mg/dL. If serum bilirubin greater than 2 mg/dl and direct bilirubin is less than 30 percent of total bilirubin contact study chair for eligibility exception for Gilbert's syndrome.
   3. ALT/AST less than or equal to 3 times the upper limit of normal
   4. LVEF 50 percent by echocardiogram or MUGA
7. Patients with history of second malignancies in complete remission and without history of metastasis are eligible if there is clinical evidence of disease stability for a period of greater than 6 months off cytotoxic chemotherapy, documented by imaging, tumor marker studies, etc., at screening.
8. Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 120 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
9. Women of child-bearing potential has negative pregnancy test prior to initiating study drug dosing.

Exclusion Criteria:

1. Current or anticipated use of additional investigational agents.
2. Any prior treatment for AML with the exception of corticosteroids, hydroxyurea, and/or leukapheresis to prevent or treat early complications prior to starting study therapy. Permitted prior therapy must be stopped 24 hours prior to starting study therapy.
3. Prior use of hypomethylating agents is permitted for patients with history of antecedent MDS. Last dose of hypomethylating therapy must have been 15 or more days prior to starting study therapy. Toxicities associated with prior MDS therapy must have recovered to grade 1 or less prior to start of treatment.
4. Favorable risk cytogenetics as defined by 2017 ELN risk stratification including acute promyelocytic leukemia
5. Chronic myeloid leukemia in myeloid blast crisis
6. Except for CMML, patients with history of myeloproliferative neoplasms (MPN) (defined as a history of essential thrombocytosis or polycythemia vera, or idiopathic myelofibrosis prior to the diagnosis of AML) or combined MDS/MPN are not eligible
7. Clinical evidence of active CNS leukemia
8. Active or metastatic second malignancy
9. Any major surgery or radiation therapy within four weeks.
10. Patients with prior cumulative anthracycline exposure of greater than 368 mg/m2 daunorubicin (or equivalent).
11. Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent obtaining informed consent
12. Patients with myocardial impairment of any cause (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV staging)
13. Active or uncontrolled infection. Patients with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for greater than or equal to 72 hrs.
14. Current evidence of invasive fungal infection (blood or tissue culture); patients with recent fungal infection must have subsequent negative culture(s) to be eligible
15. Known HIV infection
16. Active hepatitis B or hepatitis C infection
17. Hypersensitivity to cytarabine, daunorubicin or liposomal products
18. History of Wilson's disease or copper-metabolism disorder
19. Pregnant or breastfeeding
20. Any condition which in the opinion of the investigator will interfere with the ability of the subject to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate after induction | 35 days
  Overall response rate after induction, defined as the sum of complete response (CR) rate and complete response with incomplete count recovery (CRi) rate after 1-2 cycles of induction therapy, in accordance with 2017 ELN criteria.

SECONDARY OUTCOMES:
Safety and Tolerability | 6 months
  Safety and tolerability will be determined by rates of NCI CTCAE 5.0 Grade 3-5 toxicities and rate of discontinuation from study therapy due to intolerance
Incidence of Grade 3 Treatment Emergent Adverse Events [Safety and Tolerability] | 6 months
  Safety and tolerability will be determined by rates of NCI CTCAE 5.0 Grade 3 toxicities and rate of discontinuation from study therapy due to intolerance
Incidence of Grade 4 Treatment Emergent Adverse Events [Safety and Tolerability] | 6 months
  Safety and tolerability will be determined by rates of NCI CTCAE 5.0 Grade 4 toxicities and rate of discontinuation from study therapy due to intolerance
Incidence of Grade 5 Treatment Emergent Adverse Events [Safety and Tolerability] | 6 months
  Safety and tolerability will be determined by rates of NCI CTCAE 5.0 Grade 5 toxicities and rate of discontinuation from study therapy due to intolerance
CR Rate | 60 days
  CR rate defined as proportion of patients achieving a CR after 1-2 cycles of induction
Overall response rate | 35 days
  Overall response rate (CR +CRi) after 1 cycle of induction
Overall survival | 1 year
  Overall survival (OS) at 1 year, with OS defined as time from start of study therapy to death from any cause
Overall survival | 3 years
  Overall survival (OS) at 3 years, with OS defined as time from start of study therapy to death from any cause
Leukemia-free survival | 1 years
  Leukemia-free survival (LFS) at 1 year, with EFS defined as the time from start of study therapy until failure to attain CR, relapse, or death from any cause
Leukemia-free survival | 3 years
  Leukemia-free survival (LFS) at 3 years, with EFS defined as the time from start of study therapy until failure to attain CR, relapse, or death from any cause
Event free survival | 1 year
  Event Free Survival (EFS) at 1 year, with EFS defined as the time from start of study therapy until failure to attain CR, relapse, or death from any cause.
Event free survival | 3 years
  Event Free Survival (EFS) at 3 years, with EFS defined as the time from start of study therapy until failure to attain CR, relapse, or death from any cause.
Platelet Recovery | 60 days
  Platelet recovery, defined as the time from start of study therapy until absolute neutrophil count >1,000/mcl in patients achieving a CR
30-day | 30 days from start of study therapy
  30-day mortality defined as death from any cause within 30 days of starting study therapy
60-day mortality | 60 days from start of study therapy
  60-day mortality defined as death from any cause within 60 days of starting study therapy

OTHER OUTCOMES:
Minimal Residual Disease (MRD) Response (positive or negative) | 60 days
  MRD response at CR/CRi will be assessed by multiparameter flow cytometry at the University of Washington.
Descriptive Statistics of Patients Mutation Profile at Screening | At Screening
  Somatic mutation profile as determined by next generation sequencing will be performed for recurrent AML mutations using standard technique used at individual sites (local or send-out testing)
Descriptive Statistics of Patients Mutation Profile at Relapse | At Relapse
  Somatic mutation profile as determined by next generation sequencing will be performed for recurrent AML mutations using standard technique.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Wieduwilt, MD, PhD, Study Chair — UC San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States